CLINICAL TRIAL: NCT03130114
Title: Antibiotics for Children With Severe Diarrhoea
Acronym: ABCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Center for Public Health Kinetics (Other); Kenya Medical Research Institute (Other); University of Washington (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); University of Liverpool (Other); Centre pour le developpement des vaccines, Mali (Unknown); University of Maryland, College Park (Other); Aga Khan University (Other); Muhimbili University of Health and Allied Sciences (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ayesha De Costa, Scientist, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC.0002722
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Diarrhea
Keywords: Mortality; Infant; Antibiotics; Linear Growth
MeSH Terms: conditions — Diarrhea | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug (azithromycin) will be delivered as dry powder, in opaque glass bottles. Control children with receive placebo powder that will appear, smell, and taste similar to the active drug. All drug bottles will be coded with participant numbers only, so that no-one will know the contents of the bottle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Placebo mixture, 0.25 ml / kg / day
  Interventions: Other: Placebo
- Azithromycin (Experimental): Azithromycin mixture (40 mg / ml), 0.25 ml / kg / day
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Participants will receive rehydration, dietary counseling, one 20 mg tablet of zinc per day and 10 mg (0.35 ml) / kg of azithromycin syrup per day, for three days
  Arms: Azithromycin
Other: Placebo — Participants will receive rehydration, dietary counseling, one 20 mg tablet of zinc per day and 0.25 ml / kg of placebo drug syrup per day, for three days
  Arms: Control

SUMMARY:
Although the current World Health Organization (WHO) recommended management package for acute diarrhoea (ORS, zinc and feeding advice) has contributed to significant reductions in diarrhoea associated mortality, over half a million children continue to die annually as a result of acute diarrhoeal episodes. In addition, rates of mortality in young children in the 90 days following an episode of acute diarrhoea appear at least as high as mortality that occurs during the acute episode. The long-term benefits of antibiotic administration may result from direct antimicrobial effects on pathogens or from other incompletely understood mechanisms including improved nutrition, alterations in immune tolerance or improved enteric function. Optimizing antibiotic treatment of acute diarrhoea episodes in very young children with severe disease may offer the opportunity to significantly reduce diarrhoea associated deaths in the 180 days following presentation for acute diarrhoea and may also improve growth.

The investigators propose to evaluate the efficacy of an antibiotic (azithromycin) delivered in a specific, targeted fashion to young children (< 2 years of age) at high risk of diarrhoea associated mortality in a multi-site randomized, double-blind, placebo-controlled trial. The study will evaluate the ability of the intervention to reduce mortality within 180 days of the acute diarrhoeal episode, and improve nutritional status over the first 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 - 23 months, presenting to a designated health care facility at a participating study site with
* Diarrhoea per caregiver perception and at least 3 loose or watery stools in the previous 24 hours,
* Diarrhoea for less than 14 days prior to screening and with at least one of the following criteria at presentation:

  * Signs of some or severe dehydration as per WHO Pocket Book 2013
  * Moderately wasted as defined by a mid-upper arm circumference (MUAC) less than 125 mm (but greater than or equal to 115 mm) or a weight-for-length z-score (WLZ) greater than -3 standard deviations (SD) and less than or equal to -2 SD after rehydration during stabilization period or
  * Severely stunted (length-for-age z-score (LAZ) <-3 SD) and
* Parent or guardian (caregiver) willing to allow household visits on day 2 and day 3 and willing to return to facility on day 90 and
* Parent or guardian (caregiver) provides a consent for trial participation on behalf of the child, based on local standards

Exclusion Criteria:

* Dysentery (gross blood in stool reported by caregiver or observed by healthcare worker (HCW)),
* Suspected Vibrio cholerae infection (determined according to WHO guidelines or clinical suspicion),
* Previously or currently enrolled in the ABCD study,
* Concurrently enrolled in another interventional clinical trial,
* Sibling or other child in the household enrolled in the ABCD study and currently taking study medication,
* Signs of associated infections (pneumonia, severe febrile illness, meningitis, mastoiditis or acute ear infection) requiring antibiotic treatment,
* Documented antibiotic use in the 14 days prior to screening (not including standard use of prophylactic antibiotics, i.e. co-trimoxazole use in human immunodeficiency virus (HIV) -exposed children),
* Documented use of metronidazole within the last 14-days,
* Known allergy or contraindication to azithromycin antibiotics,
* Severe acute malnutrition (SAM) defined as weigh-for-length Z-score (WLZ) less than -3 SD, or MUAC less than 115 mm, or edema of both feet, or
* Living too far from the enrolment health center to ensure adequate Directly Observed Therapy (DOT) on day 2 and day 3

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8268 (Actual)
Dates: Start 2017-05-13 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 180 days from enrolment
  Proportion of children dying per arm
Linear growth | 90 days from enrolment
  Mean change in length-for-age Z-score per arm. The Z score will be arrived at from the WHO growth charts based on length in cms and age in months

SECONDARY OUTCOMES:
Hospitalizations upto Day 90 | 90 days
  Proportion of children with at least one hospitalization upto Day 90 per arm
Hospitalization or deaths upto day 90 | 90 days
  Proportion of children with at least one hospitalization or death upto day 90 per arm
Early hospitalization or death (upto day 10) | 10 days
  Proportion of children with death or any hospitalization per arm (upto day 10)
Change in weight for length Z score | 90 days
  Mean change in weight-for-length Z-score per arm. The Z score will be arrived at from the WHO growth charts based on weight in kg and length in cm for each child
Change in weight for age Z score | 90 days
  Mean change in weight-for-age Z-score per arm. The Z score will be arrived at from the WHO growth charts based on weight in kg and age in months for each child
Change in Mid upper arm circumference | 90 days
  Mean change in MUAC (mm) per arm
Antimicrobial resistance in the community | Baseline
  Proportion of study participants per arm harbouring antibiotic resistant E. coli bacteria in their stools before any intervention
Antimicrobial resistance among the study participants (sub-group) | At the end of intervention (90 days) and three months later (180 days)
  Proportion of study participants per arm harbouring antibiotic resistant S. pneumoniae bacteria in the naso-pharynx or E. coli bacteria in their stools
Antimicrobial resistance among close household child contacts (sub-group) | At the end of intervention (90 days) and three months later (180 days)
  Proportion of siblings or other close household contacts (6-59 months old) per arm harbouring antibiotic resistant S. pneumoniae bacteria in the nasopharynx or E. coli bacteria in their stools

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Bahl, Study Director — World Health Organization
Locations (7):
- Icddr,B, Dhaka, Bangladesh
- Centre for Public Health Kinetics, New Delhi, India
- Kenya Medical Research Institute, Nairobi, Kenya
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi
- Centre pour le Développement des Vaccins (CVD-Mali), Bamako, Mali
- Aga Khan University, Karachi, Pakistan
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided
The Principal investigators are currently discussing this between themselves and their research organizations. The plan is to make the data available as soon as possible.

REFERENCES:
- [Derived] Somji S, Ashorn P, Manji K, Ahmed T, Chisti M, Dhingra U, Sazawal S, Singa B, Walson JL, Pavlinac P, Bar-Zeev N, Houpt E, Dube Q, Kotloff K, Sow S, Yousafzai MT, Qamar F, Bahl R, De Costa A, Simon J, Sudfeld CR, Duggan CP; ABCD Study Group. Clinical and nutritional correlates of bacterial diarrhoea aetiology in young children: a secondary cross-sectional analysis of the ABCD trial. BMJ Paediatr Open. 2024 Apr 11;8(1):e002448. doi: 10.1136/bmjpo-2023-002448. PMID 38604769
- [Derived] Pavlinac PB, Platts-Mills JA, Liu J, Atlas HE, Gratz J, Operario D, Rogawski McQuade ET, Ahmed D, Ahmed T, Alam T, Ashorn P, Badji H, Bahl R, Bar-Zeev N, Chisti MJ, Cornick J, Chauhan A, De Costa A, Deb S, Dhingra U, Dube Q, Duggan CP, Freyne B, Gumbi W, Hotwani A, Kabir M, Islam O, Kabir F, Kasumba I, Kibwana U, Kotloff KL, Khan SS, Maiden V, Manji K, Mehta A, Ndeketa L, Praharaj I, Qamar FN, Sazawal S, Simon J, Singa BO, Somji S, Sow SO, Tapia MD, Tigoi C, Toure A, Walson JL, Yousafzai MT, Houpt ER; AntiBiotics for Children with severe Diarrhea (ABCD) Study Group. Azithromycin for Bacterial Watery Diarrhea: A Reanalysis of the AntiBiotics for Children With Severe Diarrhea (ABCD) Trial Incorporating Molecular Diagnostics. J Infect Dis. 2024 Apr 12;229(4):988-998. doi: 10.1093/infdis/jiad252. PMID 37405406
- [Derived] Antibiotics for Children With Diarrhea (ABCD) Study Group; Ahmed T, Chisti MJ, Rahman MW, Alam T, Ahmed D, Parvin I, Kabir MF, Sazawal S, Dhingra P, Dutta A, Deb S, Chouhan A, Sharma AK, Jaiswal VK, Dhingra U, Walson JL, Singa BO, Pavlinac PB, McGrath CJ, Nyabinda C, Deichsel EL, Anyango M, Kariuki KM, Rwigi D, Tornberg-Belanger SN, Kotloff KL, Sow SO, Tapia MD, Haidara FC, Mehta A, Coulibaly F, Badji H, Permala-Booth J, Tennant SM, Malle D, Bar-Zeev N, Dube Q, Freyne B, Cunliffe N, Ndeketa L, Witte D, Ndamala C, Cornick J, Qamar FN, Yousafzai MT, Qureshi S, Shakoor S, Thobani R, Hotwani A, Kabir F, Mohammed J, Manji K, Duggan CP, Kisenge R, Sudfeld CR, Kibwana U, Somji S, Bakari M, Msemwa C, Samma A, Bahl R, De Costa A, Simon J, Ashorn P. Effect of 3 Days of Oral Azithromycin on Young Children With Acute Diarrhea in Low-Resource Settings: A Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2136726. doi: 10.1001/jamanetworkopen.2021.36726. PMID 34913980
- [Derived] ABCD study team. A double-blind placebo-controlled trial of azithromycin to reduce mortality and improve growth in high-risk young children with non-bloody diarrhoea in low resource settings: the Antibiotics for Children with Diarrhoea (ABCD) trial protocol. Trials. 2020 Jan 13;21(1):71. doi: 10.1186/s13063-019-3829-y. PMID 31931848

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03130114/SAP_000.pdf
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT03130114/Prot_001.pdf